CLINICAL TRIAL: NCT01211860
Title: A Multiple-Dose Pharmacokinetic Study of Diazoxide Choline Controlled-Release Tablet (DCCR) in Subjects With Elevated Fasting Triglyceride Levels
Brief Title: Pharmacokinetic Study of Diazoxide Choline in Hypertriglyeridemic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Essentialis, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PK015
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hypertriglyceridmia
Keywords: DCCR; Diazoxide Chonline Controlled-Release Tablet = DCCR; Hypertriglyceridemia; Triglycerides; Pharmacokinetics
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCCR Treatment (Experimental): DCCR Treatment 290 mg diazoxide choline
  Interventions: Drug: Diazoxide Choline Controlled-Release Tablet

INTERVENTIONS:
Drug: Diazoxide Choline Controlled-Release Tablet — DCCR 290 mg once a day for 10 days

SUMMARY:
Once a day oral administration with DCCR is the optimal dosing regimen

DETAILED DESCRIPTION:
POPULATION The population will consist of generally healthy subjects with elevated fasting triglyceride levels in the range of ≥ 150 mg/dL and ≤ 1500 mg/dL at the Screening Visit.

Number of Subjects A total of 10 subjects will be enrolled in the study at 1 site in the USA.

ELIGIBILITY:
Inclusion Criteria:

Basic requirements

1. Healthy male and female subjects 18 to 75 years of age, inclusive at the time of dosing
2. Body mass index (BMI) between 22 and 35 kg/m2

   Specific laboratory test results
3. Fasting triglyceride ≥ 150 mg/dL and ≤ 1500 mg/dL
4. Fasting glucose ≤ 110 mg/dL
5. HbA1c ≤ 6.0 %

Exclusion Criteria:

Medications: recent, current, anticipated

1. Thyroid hormones or preparations within 1 month prior to Screening Visit (except in subjects on stable dose of replacement therapy for at least 1 month)
2. Thiazide diuretics within 2 weeks prior to Screening Visit

   History of allergic reaction or significant intolerance to:
3. Diazoxide
4. Thiazides
5. Sulfonamides

   Lifestyle changes
6. Subjects intending to change exercise habits, and/or quit smoking

   Specific diagnoses, medical conditions and history
7. Known type I or III hyperlipidemia
8. Known type 1 DM
9. Known type 2 DM
10. Any other clinically significant endocrine, cardiovascular, pulmonary, neurological, psychiatric, hepatic, gastrointestinal, hematological, renal, or dermatological disease interfering with the assessments of the investigational drug, according to the Investigator

    Specific laboratory test results
11. Any relevant biochemical abnormality interfering with the assessments of the investigational drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Steady-state Pharmacokinetic profile of DCCR | 10 days
  * Mean concentration-time profile for diazoxide
  * Steady-state pharmacokinetic parameters of diazoxide (Cmax(ss), AUC0-inf(ss), and CL/F)
  * Terminal elimination half-life (t½) of diazoxide

SECONDARY OUTCOMES:
Concentration-Time profile of major metabolite | 10 days
  * Steady-state pharmacokinetic parameters (Cmax(ss) and AUC0-inf(ss)) of the major metabolite of diazoxide
  * Terminal elimination half-life (t½) of the major metabolite of diazoxide
  * Metabolite-to-parent ratios at steady-state in terms of Cmax(ss) and AUC0-inf(ss)

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Copa, PharmD, Principal Investigator — Cetero Research - Fargo, ND
Locations (1):
- Cetero, Fargo, North Dakota, United States